CLINICAL TRIAL: NCT01533545
Title: Effect of Epinephrine on Systemic Absorption of Mepivacaine Administered for Brachial Plexus Block in Patients With Chronic Renal Insufficiency
Brief Title: Effect of Epinephrine on Systemic Absorption of Mepivacaine in Uremic Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Robertas Martusevicius, Principal Investigator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-3-2011-154; 2012-000948-98 (EudraCT Number)
Record Dates: First submitted 2012-02-08; First posted 2012-02-15 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2014-04

CONDITIONS: Renal Insufficiency, Chronic
Keywords: Mepivacaine; Epinephrine; Brachial plexus block; Renal insufficiency
MeSH Terms: conditions — Renal Insufficiency, Chronic; Renal Insufficiency | interventions — Mepivacaine; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Plain mepivacaine (Active Comparator)
  Interventions: Drug: Plain mepivacaine
- Mepivacaine with epinephrine (Active Comparator)
  Interventions: Drug: Mepivacaine with epinephrine

INTERVENTIONS:
Drug: Mepivacaine with epinephrine — Ultrasound-guided infraclavicular brachial plexus block with mepivacaine 400 mg (10 mg/mL) mixed with epinephrine 200 μg (5 μg/mL)
  Other Names: Carbocain-Adrenalin
  Arms: Mepivacaine with epinephrine
Drug: Plain mepivacaine — Ultrasound-guided infraclavicular brachial plexus block with plain mepivacaine 400 mg (10 mg/mL)
  Other Names: Carbocain
  Arms: Plain mepivacaine

SUMMARY:
The aim of this study is to determine the effect of epinephrine on systemic absorption of local anaesthetic mepivacaine administered for brachial plexus block in uremic patients scheduled for creation or repair of an arteriovenous fistula. Furthermore, an impact of epinephrine on the central circulation and peripheral tissue oxygenation will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* patient acceptance of regional anaesthesia

Exclusion Criteria:

* peripheral arteriosclerosis
* diabetes mellitus
* bleeding disorder
* infection at the puncture site
* allergy to mepivacaine
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-09; Primary Completion 2014-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Plasma concentration of mepivacaine | 0, 5, 10, 20, 30, 45, 60, 120, and 180 min after blockade

SECONDARY OUTCOMES:
Central circulation | 0, 5, 10, 15, 20, 25, 30, 35, 40, 45, 50, 55, and 60 min after blockade
  Heart rate, blood pressure, cardiac output, stroke volume, and systemic vascular resistance
Peripheral tissue oxygenation | 0, 5, 10, 15, 20, 25, 30, 35, 40, 45, 50, 55, and 60 min after blockade
  Near infrared spectrometry obtained from the triceps muscle of the blocked arm
Cardiotoxicity of local anesthetic | 0, 5, 10, 20, 30, 45, and 60 min after blockade
  12-lead ECG
Neurotoxicity of local anesthetic | Continuously for 1 hour after blockade
  Visual and hearing disturbances, dysarthria, tingling, perioral numbness, dizziness, paraesthesia, muscular twitching and rigidity

CONTACTS AND LOCATIONS:
Overall Officials: Robertas Martusevicius, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Background] McEllistrem RF, Schell J, O'Malley K, O'Toole D, Cunningham AJ. Interscalene brachial plexus blockade with lidocaine in chronic renal failure--a pharmacokinetic study. Can J Anaesth. 1989 Jan;36(1):59-63. doi: 10.1007/BF03010889. PMID 2914337
- [Background] Norio K, Makisalo H, Isoniemi H, Groop PH, Pere P, Lindgren L. Are diabetic patients in danger at renal transplantation? An invasive perioperative study. Eur J Anaesthesiol. 2000 Dec;17(12):729-36. doi: 10.1046/j.1365-2346.2000.00760.x. PMID 11122310
- [Background] Niemi G. Advantages and disadvantages of adrenaline in regional anaesthesia. Best Pract Res Clin Anaesthesiol. 2005 Jun;19(2):229-45. doi: 10.1016/j.bpa.2004.12.004. PMID 15966495
- [Background] Rosenberg PH, Veering BT, Urmey WF. Maximum recommended doses of local anesthetics: a multifactorial concept. Reg Anesth Pain Med. 2004 Nov-Dec;29(6):564-75; discussion 524. doi: 10.1016/j.rapm.2004.08.003. PMID 15635516